CLINICAL TRIAL: NCT04198792
Title: Predictors for Survival and Good Neurological Outcome in E-CPR and Non CPR Treated Patients
Status: Recruiting | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Bengt Redfors, MD, PhD, Associate Professor, Sahlgrenska University Hospital
Other Study IDs: GES
Record Dates: First submitted 2019-11-18; First posted 2019-12-13 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Cardiac Arrest; Extracorporeal Membrane Oxygenation; Hypoxia-Ischemia, Brain
MeSH Terms: conditions — Heart Arrest; Hypoxia-Ischemia, Brain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ECPR patients: Patients that is put om ECMO during cardiac arrest
  Interventions: Other: No intervention
- ECMO patients, non-ECPR: Patients that is put on ECMO due to circulatory failure but not cardiac arrest
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention, but ECPR patients will be compared to ECMO-patients that have not had cardiac arrest

SUMMARY:
In ECPR, where CPR times often range from 30 to 120 minutes, only patients with good circulation during CPR survive, while non-survivors commonly suffer from anoxic brain injury. The selection process during CPR is challenging causing a general survival rate of just 2 out of 10, and the urgent need for better selection criteria has been emphasized. It it crucial to keep cardiac arrest times as short as possible, pre primed-ECMO can facilitate this.

The ECMO treatment and the long CPR times of ECPR can also affect the measurements of the neurologic prognostication guidelines after cardiac arrest, making its validity uncertain in this specific cohort. Further, the long-term neuropsychological follow-up is limited to a few patients, making it uncertain if ECPR gives the survivors good long-term life satisfaction or just a prolonged life.

Our overall aim is to optimize and improve the care pathway for ECPR patients by refining patient selection, assessing pre-primed ECMO, validating neurological prognostication guidelines, and understanding long-term outcomes and challenges faced by survivors.

Specific Aim 1: Evaluating predictors for good neurological outcomes in ECPR and to develop and validate (internally and externally) an evidence-based selection tool for ECPR.

Specific aim 2: To assess the sterility and function of pre-primed ECMO.

Specific aim 3: To evaluate the applicability of current guidelines for neurological prognostication after cardiac arrest in ECPR patients, and to assess the predictive value of individual and combined neurological tests in this specific patient population.

Specific aim 4: To determine the long-term neuropsychological outcomes, identify the problems survivors experience in daily life, and assess life satisfaction - by comprehensive follow-up visits with validated questionnaires and neuropsychology testing up to 12 years after the ECMO-treated cardiac arrest.

DETAILED DESCRIPTION:
Specific aim 1: The aim is to develop an ECPR prognostication tool and validate its performance. In development, possible predictors for good neurological outcomes are prospectively gathered. The predictive ability of the predictors is tested in univariate and multivariable analysis, with the aim of improving patient selection for ECPR. Patients from the Gothenburg ECPR cohort are included in the development study. External validation with the ECMO patients from the Prague OHCA trial, following guidelines for validation studies, will follow, as well as external validation with further patients from Gothenburg.

Specific aim 2: Cardiohelp ECMO circuits are set up dry, followed by wet-priming and used in the ECMO treatments of the centre. The circuits are cultured at ECMO-initiation and the incidence of positive cultures is assessed. The effect of the pre-primed time on ECMO function is also assessed.

Specific aim 3: The predictive ability of the current guideline for neurological prognostication of comatose patients in the ICU after cardiac arrest, from the European Resuscitation Council, is assessed in the ECPR cohort of Gothenburg. The diagnostic performance of individual predictors as well as the total accuracy of the prediction will be assessed.

Specific aim 4: A Long-term (1-12 years) follow-up of the ECPR patients will be performed, to determine the long-term neuropsychological outcomes.

4 A: Life satisfaction after ECPR will be assessed along with anxiety, depression, fatigue, cognitive function, and physical activity. The impact of these factors on life satisfaction will also be evaluated. QUALY will be calculated.

4 B: Long-term neurocognitive function in ECPR patients will be assessed through comprehensive neuropsychological testing, using conventional CPR patients from the TTM2 trial as a control group.

The general ECMO population from 2004 of the center is included as a control group and positive cultures during their ECMO runs are documented.

ELIGIBILITY:
Inclusion Criteria:

* ECMO-treated patients.

Exclusion Criteria:

* None

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ECPR Group: Patients who is put on ECMO during cardiac arrest. ECMO Group: Patients who is put on ECMO with some ongoing circulaiton
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin scale (MRs) | 1 year
  Assessmenty of cognitive function. 0-6, where 0 is best.
Performance of ECMO oxygenator function | 0-60 days
  Oxygenator resistance, and the needed FiO2 and sweep gas flow will be assessed
Positive cultures of pre-primed ECMO circuits | 0-90 days
  ECMO circuits is pre-primed and cultures taken at the start of ECMO treatment
Predictive ability of ERC neuro prognostication guidelines on ECPR patients | 1 year
  Diagnostic performance and ROC analysis of individual and total ERC predictors on outcome in ECPR
Life Satisfaction | 1-12 years
  Visual Analog Scale 1-10. 10 is better.
Euro Qualy - 5 dimension (EQ-5D-5L) VAS | 3 months to 12 years
  Self-perceived health status. 0-100, where higher is better.
Neurocognitive function | 3 months to 12 years after the ECPR-treatment
  Z-scores of verbal and visual function, episodic and visuospatial memory , processing speed and executive functions. 0 represents standardized population norm and ± 1 represent one standard deviation from that.
Positive blood Cultures | 1 month
  Infection rates in ECMO-patients

SECONDARY OUTCOMES:
MoCA | 3 months to 12 years after the ECPR treatment
  Assess cognitive function, higher is better. 0-30 where higher is better
Hospital Anxiety and Depression Scale (HADS) | 3 months to 12 years
  Two sub scales 0-21 which assess anxiety and depression, higer is worse
Mental Fatigue Scale | 3 months to 12 years
  Assess fatigue 0-42 points. Higher is worse
modified Rankin Scale | 3 months to 12 years
  physical function from 0-6 where 0 is best
Actual physical activity | 3 months to 12 years
  Days per seven days with more than 30 minutes of physical activity

OTHER OUTCOMES:
Cost | 3 month
  The in hospital cost of the treatment for the patients, in Swedish kronor.
Short Form -36 (SF-36) | 1-7 years
  Quality of life. 8 scaled scores from 0-100, where 100 is best.
Trailmaking test | 1-7 years
  Assessmenty of cognitive function. Shorter time is better.
New York heart association class (NYHA class) | 1-7 years
  Assessment of physical function.1-4, where 1 is best
Euro-Qualy-5D-5L | 3 moths to 12 years
  Quality of life assessment, higher is better. Swedish value set -0.33 - 1.00

CONTACTS AND LOCATIONS:
Overall Officials: Bengt Redfors, MD, PhD, Principal Investigator — The Sahlgrenska Academy ar Sahlgrenska University Hospital, Gorhenburg, Sweden
Locations (1):
- Sahlgrenska Academy at Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bengtsson D, Jonsson B, Redfors B. Sterility and oxygenator function in pre-primed extracorporeal membrane oxygenation: A prospective clinical study. Resusc Plus. 2024 Jun 5;19:100680. doi: 10.1016/j.resplu.2024.100680. eCollection 2024 Sep. PMID 38912528
- [Result] Redfors B, Byttner A, Bengtsson D, Watson P, Lannemyr L, Lundgren P, Gabel J, Rawshani A, Henningsson A. The Pre-ECPR Score: Developing and Validating a Multivariable Prediction Model for Favorable Neurological Outcomes in Patients Undergoing Extracorporeal Cardiopulmonary Resuscitation. J Cardiothorac Vasc Anesth. 2024 Dec;38(12):3018-3028. doi: 10.1053/j.jvca.2024.09.009. Epub 2024 Sep 17. PMID 39395854